CLINICAL TRIAL: NCT07074756
Title: Neuro-Oncology Anywhere: Glioma Home-Based Sequential Therapy (GHoST) Protocol
Brief Title: A Digital Treatment Platform for the Delivery of Home-Based Sequential Therapy in Patients With Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240703; NCI-2025-04495 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-009234 (Other: Mayo Clinic Institutional Review Board); MC240703 (Other: Mayo Clinic)
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Glioma; Recurrent Glioma
MeSH Terms: conditions — Glioma | interventions — Drug Therapy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (remote chemotherapy management) (Experimental): Patients receive access to the remote chemotherapy management and patient monitoring platform to watch educational videos, report when medication is taken or missed, and report any symptoms related to cancer or medication side effects on study. Patients also receive standard of care chemotherapy as assigned by their treating physician as part of the platform on study. Upon completion of standard of care chemotherapy, if there is no disease progression, patients transition to surveillance for up to 1 year. Patients who experience disease progression during treatment or surveillance may rejoin the platform and/or be assigned by their treating physician to a different chemotherapy agent as part of the platform. Patients also undergo MRI or CT throughout the study.
  Interventions: Drug: Chemotherapy; Procedure: Computed Tomography; Other: Internet-Based Intervention; Procedure: Magnetic Resonance Imaging; Procedure: Neurologic Examination; Other: Questionnaire Administration; Behavioral: Surveillance

INTERVENTIONS:
Drug: Chemotherapy — Receive standard of care chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Internet-Based Intervention — Receive access to the remote chemotherapy management and patient monitoring platform
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Neurologic Examination — Ancillary studies
  Other Names: Nervous System Examination; Neurological Assessment; neurological exam; Neurological Examination; NVEXAM
Other: Questionnaire Administration — Ancillary studies
Behavioral: Surveillance — Undergo surveillance
  Other Names: Epidemiology / Surveillance

SUMMARY:
This clinical trial tests how well a digital treatment platform using a mobile application works for the delivery of home-based sequential therapy in patients with glioma. Access to specialized neuro-oncology care in the United States for patients with glioma is critically deficient. Care at centers with neuro-oncology specialists is associated with improved survival outcomes, yet many patients have limited access due to distance, disease-related disability, or lack of financial resources. The application provides patients continuous access to their care team in the home setting. A digital treatment platform may increase clinical trial participation and accelerate development of novel therapeutics while addressing a great health disparity in patients with glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of the remote chemotherapy management and patient monitoring platform glioma home-based sequential therapy (GHoST) protocol among patients with glioma undergoing systemic therapy.

SECONDARY OBJECTIVES:

I. Evaluate compliance, adherence, and feasibility in terms of the adherence to systemic therapy monitored remotely.

II. Determine progression free survival (PFS) for each therapeutic evaluated for newly diagnosed or recurrent glioma, stratified by tumor type.

III. Determine objective response rate (ORR) for each therapeutic evaluated for newly diagnosed or recurrent glioma, stratified by tumor type.

IV. Assess the safety and tolerability of remote chemotherapy management and patient monitoring among patients with glioma undergoing systemic therapy.

EXPLORATORY OBJECTIVES:

I. Assess the acceptance or satisfaction of patients with the remote monitoring in this trial and how these may differ between newly diagnosed and recurrent glioma.

II. Investigate PFS based on therapeutic sequence administered. III. Explore potential differences in compliance, adherence, and satisfaction measures and how they may correspond to health disparities and social determinants of health.

IV. Compare access to neuro-oncology care at Mayo Clinic among patients with low socioeconomic status assessed based on the Mayo Clinic Housing-Based Socioeconomic Status (HOUSES) Index during the two years following study activation compared to historical utilization data.

V. Compare access to neuro-oncology care at Mayo Clinic among patients with increased distance from academic centers assessed by geospatial index during the two years following study activation compared to historical utilization data.

OUTLINE:

Patients receive access to the remote chemotherapy management and patient monitoring platform to watch educational videos, report when medication is taken or missed, and report any symptoms related to cancer or medication side effects on study. Patients also receive standard of care chemotherapy as assigned by their treating physician as part of the platform on study. Upon completion of standard of care chemotherapy, if there is no disease progression, patients transition to surveillance for up to 1 year. Patients who experience disease progression during treatment or surveillance may rejoin the platform and/or be assigned by their treating physician to a different chemotherapy agent as part of the platform. Patients also undergo magnetic resonance imaging (MRI) or computed tomography (CT) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of glioma and intention to treat with either new or ongoing systemic therapy for at least 6 months.

  * NOTE: Patient may be enrolled following completion of surgery and/or radiation therapy for newly diagnosed or recurrent tumor.
  * NOTE: Any number of prior recurrences is permitted
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2, AND Karnofsky performance status (KPS) of ≥ 60
* Expected survival ≥ 6 months in the opinion of treatment team
* Willing and able to adhere with the protocol for the duration of the study including undergoing treatment, and attending scheduled visits, and examinations
* Negative pregnancy test ≤ 8 days prior to registration for persons of childbearing potential only
* Provide written informed consent
* Ability to complete assessments and questionnaires by themselves or with assistance

Exclusion Criteria:

* Pregnant or nursing, imprisoned, or lacking capacity for understanding
* Uncontrolled and/or intercurrent illness or other condition which limits safety of or compliance with study proceedings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - completion of study visits | At baseline and the set of study-specific visits through 6 months (i.e., 26 weeks ± 2 weeks)
  Feasibility will be assessed by the number of study visits completed vs. not. Will consider this to be feasible in this patient population if the true compliance rate is at least 60%. Compliance here is defined as completion of at least 4 disease assessment timepoints in the first 6 months on study (i.e. 26 ± 2 weeks). These assessment timepoints will include the baseline assessment and can include assessments after 2 cycles of therapy, after 4 cycles of therapy, after 6 cycles of therapy, dependent on the treatment-specific schedules.

SECONDARY OUTCOMES:
Acceptance of and satisfaction of patients with the remote monitoring | Up to 3 years
  Will be assessed with an electronic Assessment of Acceptance and Satisfaction survey sent to participants at study assessment timepoints. The satisfaction survey consists of a single question answered on a 5-point scale: very positive, somewhat positive, neutral, somewhat negative, very negative.
Adherence to study therapeutics | Up to 3 years
  Will be assessed through remote monitoring application. Here, adherence is defined as taking at least 80% of the prescribed doses, for all therapies other than lomustine. For lomustine, adherence is defined as receiving all prescribed infusions.
Feasibility of remote systemic therapy assessments | Up to 3 years
  Will be assessed through completion of visits as scheduled, where laboratory and imaging assessed for the visits are scheduled and completed prior to telehealth visits. Feasibility will be defined as having necessary pre-visit testing completed and delivered for clinician review prior to the visit as well as completion of the visit at the intended scheduled time for 60% of the visits.
Progression free survival (PFS) for each therapeutic treatment diagnosed and recurrent glioma | At 6 months
  Will be assessed for each treatment evaluated. PFS is defined as the time from enrollment to disease progression or death, whichever occurs first.
Objective response rate | Up to 3 years
  Objective response rate for each therapeutic for newly diagnosed and recurrent glioma will be assessed.
Incidence of adverse events | Up to 3 years
  Will be assessed by type along with grade and perceived attribution to study agent based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Safety of the overall platform | Up to 3 years
  Will be assessed by acute care utilization days (defined as emergency department evaluations and inpatient days) for participants on the platform compared to historical clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur T. Sener, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Related Info — https://www.mayo.edu/research/clinical-trials